CLINICAL TRIAL: NCT05972330
Title: Testing the Efficacy of VRx MyBiotics Oral Lozenges to Improve the Oral Microbiome
Brief Title: Efficacy of VRx MyBiotics Oral Lozenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: V308
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Oral Microbiome Health
Keywords: oral health; oral lozenge; oral microbiome

STUDY DESIGN:
Intervention Model Description: Participants will be assigned an oral lozenge formulation based on the baseline analysis of their oral microbiome.
Masking Description: None, Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRx MyBiotics Oral Lozenges (Experimental): Participants will receive a 30 day supply of their personalized oral biotic lozenges.
  Interventions: Dietary Supplement: VRx MyBiotics Oral Lozenges

INTERVENTIONS:
Dietary Supplement: VRx MyBiotics Oral Lozenges — VRx MyBiotics Oral Lozenges are composed of prebiotics, probiotics, and postbiotics.

SUMMARY:
This study will test the efficacy of Viome's VRx MyBiotics Oral Lozenges at improving the oral microbiome.

DETAILED DESCRIPTION:
This is a single arm, interventional trial on adults residing in the United States. The study will test the efficacy of personalized oral biotic lozenges (VRx MyBiotics Oral Lozenges) at improving oral microbiome health according to Viome's Oral Health Score.

ELIGIBILITY:
Inclusion Criteria:

* Any person with a US address that is 18 years old or older
* Able to speak and read English
* Willing and able to follow the trial instructions, as described in the recruitment letter
* Signed and dated informed consent prior to any trial-specific procedures.

Exclusion Criteria:

* Systemic antibiotic treatment 30 days prior to enrollment or during the trial
* Not willing to stop sporadic use (less frequently than daily) of any mouthwash.
* Significant diet, supplements, or lifestyle change in the previous 1 month or next 2 months once enrolled
* Allergy to tapioca, peppermint, or sweet potato
* Current diagnosis of periodontitis or other advanced oral disease (chronic recurrent caries, oral cancer, etc)
* No dental procedures 30 days prior to enrollment or during the trial (regular cleanings, bone grafts, dental implants, etc)
* Pregnancy or planned pregnancy
* Currently have cancer or undergoing cancer therapy
* Dentures
* Fewer than 20 teeth
* Use of at home teeth whitening products 30 days prior to enrollment or during the trial
* Start new medications or supplements during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Viome Oral Health Score | ~ 4 months
  Increase in oral health score as measured by Viome's Oral Health Score.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States